CLINICAL TRIAL: NCT04180943
Title: Liposomal Bupivacaine Versus Bupivacaine for Interscalene Nerve Block for Postoperative Pain Control in Shoulder Arthroplasty/Arthroscopy: a Prospective Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine Versus Bupivacaine for for Postoperative Pain Control in Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Linda Demma, MD, PhD, attending physician - anesthesiology, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1422773
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- liposomal bupivicaine (Active Comparator): interscalene nerve block using liposomal bupivacaine (Exaprel) 10 ml mixed with 0.5% bupivacaine in same syringe - volume of bupivacaine per MD based on pt weight, etc but CANNOT EXCEED 13mL
  Interventions: Drug: interscalene nerve block
- bupivicaine (Active Comparator): interscalene block using standard bupivicaine (combination of ropivacaine 0.5% and lidocaine 2%) (volume per MD based on pt weight) + decadron
  Interventions: Drug: interscalene nerve block

INTERVENTIONS:
Drug: interscalene nerve block — intra and post-operative analgesia
  Other Names: liposomal bupivicaine

SUMMARY:
This is a randomized, single blinded clinical trial whose purpose is to assess the impact of liposomal bupivacaine (LB) in a single shot interscalene nerve block compared with standard bupivacaine (same dose) in a single shot interscalene nerve block in terms of postoperative pain control. Specifically, outpatient pain scores,use of postoperative pain medicine and patient-reported functional outcomes after shoulder arthroplasty surgery will be evaluated.

DETAILED DESCRIPTION:
Background:

Shoulder arthroplasty is the fastest growing joint replacement surgery in the United States, and optimal postoperative pain management is critical to optimize outcomes for these surgeries. LB has gained popularity for its potential to provide extended postoperative pain relief with possibly fewer side effects. LB (Exparel, Pacira Pharmaceuticals, Inc., Parsippany, NJ, USA) has recently gained popularity for its potential to provide extended postoperative pain relief and was recently approved by the FDA for use in interscalene nerve blocks. Several studies have investigated its efficacy after hip and knee arthroplasty and demonstrated efficacy with decreased opioid consumption, early mobilization, lower hospital costs, and shorter length of stay for patients undergoing surgeries such as bunionectomy, open colectomy, umbilical hernia repair, breast augmentation, and total knee arthroplasty. Limited studies have evaluated the efficacy of LB for perioperative pain control in shoulder arthroplasty. Hence, the objective of this study is to determine whether the use of an LB-based multimodal analgesic regimen provides better postoperative pain control and patient satisfaction, greater cost effectiveness, and lower risk profile compared with standard bupivacaine in interscalene nerve bloc

Study Design and Methods:

This will be a prospective, randomized, single blinded, controlled clinical trial comparing patients undergoing shoulder arthroscopy and arthroplasty treated with LB versus standard bupivacaine with a single bolus interscalene block. The block administrator will not be blinded. The patient and the staff members conducting the follow up assessments, phone calls, and data collection will be blinded to treatment assignment. Study drug administrators (anesthesiologists) will not be blinded. There will be at least one unblinded study coordinator who will not be involved in collecting outcome data.

Patients will be randomized in 1:1 ratio to LB or standard bupivacaine with a single bolus interscalene block. Patient will receive the assigned interscalene block preoperatively per usual procedure. The primary outcome, time to first post operative pain medication will be recorded either from the medical record if administered in the hospital or via telephone assessment if consumed outside the hospital. Study staff will contact the patient by phone post op day (POD) 1, 2, and 3 to assess pain levels, pain medication consumption, sleep, and adverse events. The total participation time for each patient will be approximately four days (operative day and POD 1,2,3).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* undergoing shoulder arthroscopy or arthroplasty
* must meet the criteria for standard of care of ambulatory surgery patients per anesthesia guidelines issued by the American Society of Anesthesiologists

Exclusion criteria:

* contraindications to regional anesthesia,
* allergy to any component of multimodal analgesia
* history of opioid use of >50 morphine milligram equivalents (MME) daily,
* significant peripheral neuropathy or neurologic disorder affecting the upper extremity,
* cognitive or psychiatric condition that might affect the patient?s assessment or inability to provide informed consent
* pregnancy (this is an exclusion for surgery as well)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Time to first post-operative pain medication consumption in minutes from discharge from OR | 72 hours
  time to first post-operative pain medication

SECONDARY OUTCOMES:
Worst daily post-op pain on a scale 1-10 | 72 hours
  patient reported outcome of pain severity
Least daily post-op pain on a scale 1-10 | 72 hours
  patient reported outcome of pain severity
Average daily post-op pain on a scale 1-10 | 72 hours
  patient reported outcome of pain severity
Total opioid use in morphine equivalents in the first 72 hours post-op | 72 hours
  Total post-op opioid use

CONTACTS AND LOCATIONS:
Overall Officials: Linda Demma, MD, PhD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers outside of the study investigators.

DOCUMENTS (1):
  • Informed Consent Form (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT04180943/ICF_000.pdf